CLINICAL TRIAL: NCT04851028
Title: MusiCare: Protecting Cognitive Functions and Wellbeing Using Music Therapy & Innovative Technology With an Aging Population
Brief Title: MusiCare: Music Therapy & Innovative Technology
Acronym: MusiCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Middlesex University (Other)
Collaborators: The Dunhill Medical Trust (Other); University of Padova (Other); Vrije Universiteit Brussel (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Anthony Mangiacotti, Lecturer in Psychology; Co-PI MusiCare Project, University of West London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020 Dec 14845; DUNHILL MEDICAL TRUST (Other Grant/Funding Number: RPGF2006\241)
Record Dates: First submitted 2021-03-29; First posted 2021-04-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy Aging; Cognitive Impairment
Keywords: music therapy; aging; cognitive function; robotics
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- One2One (Experimental): 1) Weekly individual (one2one) Music Therapy intervention lasting 5 months (n=20 sessions)
  Interventions: Behavioral: Music Therapy
- Small-group (Experimental): 2) Weekly small group (max 8 people per group) Music Therapy intervention lasting 5 months (n=20 sessions)
  Interventions: Behavioral: Music Therapy
- Large group (Experimental): 3) Weekly Large group (max 8 people per group) Music Therapy intervention lasting 5 months (n=20 sessions)
  Interventions: Behavioral: Music Therapy
- Control (No Intervention): Passive control, not attending any music-related activity

INTERVENTIONS:
Behavioral: Music Therapy — Music therapy is a non-pharmacological intervention, in which music and its elements are used professionally as an intervention in medical, educational, and everyday environments with individuals, groups, families, or communities who seek to optimize their quality of life and improve their physical, social, communicative, emotional, intellectual, and spiritual health and wellbeing. This therapy has shown to provide significant benefits for individuals with cognitive decline living in care homes, enhancing social-cognitive functions and reducing behavioural symptoms (Brotons & Koger, 2000; Hsu et al., 2015; Zhang et al., 2017).
  Arms: Large group; One2One; Small-group

SUMMARY:
The number of older people living with cognitive impairment or dementia has increased the need for simple, inexpensive interventions to improve the quality of life for such individuals and their families. Policy-makers sensitive to issues associated with mental health challenges in aging have embraced social prescribing, and a wealth of research has flourished to study non-pharmacological forms of preventative intervention. Can music-therapy(MT) be one of them? Different studies demonstrated that music stimulates a range of cognitive and social functions. However, scientific studies assessing the value of MT for those who need support in later life are limited, and rigorous research is required to generate robust scientific evidence. The focus of this study is on developing novel forms of intervention for older adults who are healthy or experiencing mild-to-moderate cognitive decline, aiming at [i]understanding whether MT could be used in preventive programs to support cognitive functions, [ii]identifying the best match between types of MT and levels of cognitive decline. Moreover, recent developments of Robotic-Assistance-Technologies offer opportunities to explore how such technologies may be used to contribute to older adults wellbeing when integrated within care routines to facilitate MT delivery.

Spanning across three-studies, the investigators will examine psychosocial benefits of 5-month MT interventions (one2one, small-group MT, large-group MT) in healthy older adults and impaired older adults in care homes, compared to standard care. This latter group will receive MT afterwards. Further, researchers will investigate whether Robotic-Assistance-Technologies may enrich MT interventions and have additional benefits for the participants and translatability for community-based services.

In order to measure these effects, psychological (cognitive functions, wellbeing, quality of life) and physiological (hormonal, cardiovascular & brain activity) measures will be compared before/after the intervention.

The study will elucidate relationships between different types of MT and benefits to participants wellbeing, cognitive functions & social engagement, as well as the impact of robotic assistive technologies in public health services and social care.

DETAILED DESCRIPTION:
The following objectives are addressed:

[Oi] Identifying a consistent set of convergent measures for the reliable assessment of cognition/well-being in MT studies integrating psychological measures with biomarkers; [Oii] Implementing robust MT protocols benefitting cognitive functions/well-being in ageing individuals with varying cognitive ability; [Oiii] Comparing the outcomes of one2one/small-group/large-group MT intervention in function of participants' cognitive abilities (ranging from healthy ageing to moderate impairment); [Oiv] Devising, implementing and testing a robotic platform associated with MT to facilitate therapists/caregivers' work through novel forms of interaction with ageing individuals, and potential translatability to communities.

Our research questions/hypotheses are:

[H1] Will MT benefits healthy, mildly and moderately impaired 65+ in outcome measures? MT > standard care.

[H2] Which MT treatment (one2one/small group/large group) is more effective in function of older adults' cognitive level? Best outcomes predicted as follows: healthy 65+ with small-group MT; for mildly impaired 65+, one2one = small-group MT<large group; moderately impaired 65+ with one2one MT.

[H3] Will improvements in cognitive functions derived from MT be associated with psychophysiological biomarkers? Convergent measures will be identified linking cognitive, behavioural and physiological improvement.

[H4] What are the benefits of MT for caregivers? A reduction in participant psychiatric and depressive symptoms will correspond to caregivers' workload and stress perception decrease.

[H5] Are there benefits from enriching MT with robotic technology? Specifically, the investigators hypothesize that a) the robot will have the capability of delivering interactive music training sessions, with the support of caregivers not specialised in MT and b) the continuous monitoring provided by the robotic platform will enhance the information available to therapists/caregivers without significantly burdening them.

MusiCare aims are:

[Ai] Provide care-homes, communities and policy-makers with clear guidelines concerning the utility, suitability and cost-effectiveness of Music Therapy (MT) interventions (one2one vs small-group vs large group) as a prevention/rehabilitation method suitable for social prescribing and support for positive ageing.

[Aii] Provide music therapists with robust protocols, new tests specifically designed to work through musical tasks (Music Cognitive Test).

[Aiii] Provide scholars/practitioners with a range of objective measures to select from, depending on their needs, in order to evaluate MT interventions in ageing.

[Aiv] Explore how the assistive robotic technologies can enrich MT in care-home settings by empowering care-home staff with a new active role in assisting rehabilitative activities as well as facilitating inter-generational communication between families and ageing relatives.

[Av] Increase public awareness about healthy ageing, and arts & wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65yrs
* No significant hearing impairment that would negatively interfere with the music-based interventions
* Fluent in English
* Healthy group - MMSE ≥ 24
* Cognitive impairment: mild MMSE= 18-23, moderate MMSE= 10-17

Exclusion Criteria:

* Presence of severe motor deficits that would not allow individuals to participate in the intervention
* Having taken part in a cognitive training programme or Music Therapy programme within the last 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
General cognitive functions change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  Mini-Mental State Examination (MMSE, Folstein et al., 1975): A world standardized tool for screening general cognitive function which allows the client to be placed on a cognitive functioning scale. This test is usually used to follow the course of a disease or for monitoring the response to a specific treatment, as in this case.
Music related cognitive function change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  Music Cognitive Test (MCT, Mangiacotti, 2019; - et al., 2019b) A music-based cognitive test to measure cognitive functions typically stimulated by rehabilitative music interventions.
Attentional functions change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  TMT-A (Reitan & Wolfoson, 1985) The test assesses selective attention and psychomotor speed.
Executive and spatial-cognitive abilities change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  Tangled Figure Test (Arcara et al., 2011) The test wants to evaluate participant's ability to perform figure-background discrimination and inhibition on the answers already provided as well as to recognize the contours of the figures. Mainly it is a test of visual recognition, but it requires the ability to reorganize a complex visual pattern in order to identify an increasing number of figures. Provides information on spatial-cognitive abilities, and executive and naming difficulties.

SECONDARY OUTCOMES:
Quality of Life change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  • Quality of Life in Alzheimer's Disease (Logsdon et al., 1999); The test measure quality of life in dementia. Rating is got from both the participant and the caregiver.
Mood Index change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  • Cornell Scale for Depression in Dementia (CSDD, Alexopoulos, Abrams, Young, & Shamoian, 1988); This test is specifically designed to screen depressive symptoms in older adults with dementia and cognitive impairment. It is an interviewer-administered scale relying on information from caregivers and clinician's observations.
Neuro-psychiatric symptoms change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  • Neuro-Psychiatric Inventory (NPI, Cummings, 1994) A tool that provides information on the presence of psychopathology in people with brain disorders. The NPI was developed for people with Alzheimer's disease and other dementias, but it may be useful in the assessment of behavioural changes in other conditions.
Cognitive reserve | Baseline (i.e., time 0)
  · Cognitive Reserve Index Questionnaire (CRI-Q, Nucci, Mapelli, Mondini, 2012). A tool used to quantify, in a standardized model, cognitive reserve through an interview to the participant or to the caregiver. The questionnaire collects demographic information regarding the school curriculum, work and type of free-time activities. These three different indices (CRI-School, CRI-Work and CRI-Free Time) are then combined into a single "Index of Cognitive Reserve". This test is useful in the research setting to balance study groups, as occur this project.
Wellbeing of Older People scale | Baseline vs. post- intervention period (time 0/+5-months)
  (WOOP; Hackert et al., 2020) Used as a general index of wellbeing, the scale asks participants to rate nine factors (physical health, mental health, social contacts, support, acceptance and resilience, feeling useful, independence, financial security, and living situation) according to their importance for overall wellbeing. Higher scores reflect greater self-perceived wellbeing
Sleep Quality Index | Baseline vs. post- intervention period (time 0/+5-months)
  Measured with the Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989) to assess overall sleep quality. This self-report questionnaire comprises seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction."

OTHER OUTCOMES:
Salivary Hormones index (cortisol/DHEA ratio) change from baseline/post (i.e., time 0/+5 months) | Baseline vs. post- intervention period (time 0/+5-months)
  Two types of salivary hormones will be collected: 1) Cortisol, which is associated with emotional distress and depressive symptoms (Biggio, Mostallino 2013); 2) DHEA is an age-related hormone involved in different physiological mechanisms (anti-oxidant, anti-inflammatory). The cortisol/DHEA ratio can be considered a reliable stress index.The average of three daily collections will be performed to obtain a single daily value. Three passive-drool samples are collected in a single day for each participant:
  * Before lunchtime (11.00am to 12.30am);
  * Before dinner (4pm to 5pm);
  * Evening (from 7pm to 8pm).
Salivary Hormones index (cortisol/DHEA ratio) change from baseline/mid-intervention(i.e., time 0/+10 weeks) | Baseline vs. mid-intervention period (time 0/+10 weeks)
  Two types of salivary hormones will be collected: 1) Cortisol, which is associated with emotional distress and depressive symptoms (Biggio, Mostallino 2013); 2) DHEA is an age-related hormone involved in different physiological mechanisms (anti-oxidant, anti-inflammatory). The cortisol/DHEA ratio can be considered a reliable stress index.The average of three daily collections will be performed to obtain a single daily value. Three passive-drool samples are collected in a single day for each participant:
  * Before lunchtime (11.00am to 12.30am);
  * Before dinner (4pm to 5pm);
  * Evening (from 7pm to 8pm).
Salivary Hormones index (cortisol/DHEA ratio) change from mid-/post-intervention (i.e., 10weeks/5 months) | Mid-intervention period (10 weeks) vs. post-intervention (5 months)
  Two types of salivary hormones will be collected: 1) Cortisol, which is associated with emotional distress and depressive symptoms (Biggio, Mostallino 2013); 2) DHEA is an age-related hormone involved in different physiological mechanisms (anti-oxidant, anti-inflammatory). The cortisol/DHEA ratio can be considered a reliable stress index.The average of three daily collections will be performed to obtain a single daily value. Three passive-drool samples are collected in a single day for each participant:
  * Before lunchtime (11.00am to 12.30am);
  * Before dinner (4pm to 5pm);
  * Evening (from 7pm to 8pm).
RSA change from baseline/post (i.e., time 0/+5 months) | Baseline and post- intervention period (time 0/+5-months)
  • Respiratory sinus arrhythmia (RSA): 5 min resting state
EEG change from baseline/post (i.e., time 0/+5 months) | Baseline and post- intervention period (time 0/+5-months)
  • Neural tracking of natural speech and musical sound: EEG measures of cortical activity (Di Liberto et al., 2015, 2020) - 8 electrodes, 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mangiacotti, PhD, Study Director — Middlesex University
Locations (1):
- MHA Methodist Homes, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset will be created with all the cognitive and physiological data collected from participants that will give consent to share their anonymised data.
Supporting Information: Study Protocol, SAP
Time Frame: August 2025
Access Criteria: Middlesex University FigShare

REFERENCES:
- [Background] Brotons M, Koger SM. The impact of music therapy on language functioning in dementia. J Music Ther. 2000 Fall;37(3):183-95. doi: 10.1093/jmt/37.3.183. PMID 10990596
- [Background] Hsu MH, Flowerdew R, Parker M, Fachner J, Odell-Miller H. Individual music therapy for managing neuropsychiatric symptoms for people with dementia and their carers: a cluster randomised controlled feasibility study. BMC Geriatr. 2015 Jul 18;15:84. doi: 10.1186/s12877-015-0082-4. PMID 26183582
- [Background] Zhang Y, Cai J, An L, Hui F, Ren T, Ma H, Zhao Q. Does music therapy enhance behavioral and cognitive function in elderly dementia patients? A systematic review and meta-analysis. Ageing Res Rev. 2017 May;35:1-11. doi: 10.1016/j.arr.2016.12.003. Epub 2016 Dec 23. PMID 28025173
- [Background] Folstein MF, Robins LN, Helzer JE. The Mini-Mental State Examination. Arch Gen Psychiatry. 1983 Jul;40(7):812. doi: 10.1001/archpsyc.1983.01790060110016. No abstract available. PMID 6860082
- [Background] Nucci M, Mapelli D, Mondini S. Cognitive Reserve Index questionnaire (CRIq): a new instrument for measuring cognitive reserve. Aging Clin Exp Res. 2012 Jun;24(3):218-26. doi: 10.3275/7800. Epub 2011 Jun 20. PMID 21691143
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Di Liberto GM, O'Sullivan JA, Lalor EC. Low-Frequency Cortical Entrainment to Speech Reflects Phoneme-Level Processing. Curr Biol. 2015 Oct 5;25(19):2457-65. doi: 10.1016/j.cub.2015.08.030. Epub 2015 Sep 24. PMID 26412129
- [Background] Di Liberto GM, Pelofi C, Bianco R, Patel P, Mehta AD, Herrero JL, de Cheveigne A, Shamma S, Mesgarani N. Cortical encoding of melodic expectations in human temporal cortex. Elife. 2020 Mar 3;9:e51784. doi: 10.7554/eLife.51784. PMID 32122465
- [Background] Biggio, G. and Mostallino, M.C., 2013. Stress, cortisol, neuronal plasticity, and depressive disorder. Journal of Psychopathology, 19, pp.77-83.
- [Background] Logsdon, R.G., Gibbons, L.E., McCurry, S.M. and Teri, L., 1999. Quality of life in Alzheimer's disease: patient and caregiver reports. Journal of Mental health and Aging, 5, pp.21-32.
- [Background] Arcara, G., Bisiacchi, P. S., Mapelli, D., Mondini, S., & Vestri, A. 2011. Esame Neuropsicologico Breve (ENB-2): una batteria di test per lo screening neuropsicologico, Raffaello Cortina Editore, Milano.
- [Background] Reitan, R. M., & Wolfson, D. (2009). The Halstead-Reitan neuropsychological test battery for adults-theoretical, methodological, and validational bases. Neuropsychological assessment of neuropsychiatric and neuromedical disorders, 1, 3-24.
- [Background] Mangiacotti, A., Cipriani, G., Ward, E., Franco, F. and Biasutti, M., 2019b. The Music Cognitive Test: A new music-based cognitive test. Alzheimer's & Dementia: The Journal of the Alzheimer's Association, 15(7), pp.446-P447.
- [Background] Mangiacotti, A., Hsu, M.H., Barone, C., Di Liberto, G., Van Puyvelde, M., Biasutti, M. and Franco, F., 2019a. Effects of music therapy in elderly care: cognition, biomarkers, mood and social behaviour. Alzheimer's & Dementia: The Journal of the Alzheimer's Association, 15(7), p.1144.
- [Background] Mangiacotti, A., PhD Thesis, "The Music Cognitive Test validation, training and applicability of a music-based cognitive tool for music therapists - an interdisciplinary study" University of Padua (submitted October 2019 - Viva passed 9th March 2020).